CLINICAL TRIAL: NCT00864721
Title: Phase II Trial of Sunitinib Malate in Previously Untreated NSCLC Patients Over the Age of 70
Brief Title: Sunitinib Non Small Cell Lung Cancer Patients Over 70
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-135; GA6181UU (Other: Pfizer)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Untreated NSCLC in patients > 70
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (Experimental): Sunitinib malate (Sutent) will be taken on an outpatient basis. Sunitinib malate (Sutent) should be taken at the dose of 37.5 mg/day by mouth; drug will only be taken Days 1-42 of each 42-day cycle.
  Interventions: Drug: Sutent

INTERVENTIONS:
Drug: Sutent — Sunitinib malate (Sutent) will be taken on an outpatient basis. Sunitinib malate (Sutent) should be taken at the dose of 37.5 mg/day by mouth; drug will only be taken Days 1-42 of each 42-day cycle.
  Other Names: sunitinib malate

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) sunitinib has on patients and their NSCLC.

DETAILED DESCRIPTION:
In this trial, the activity and tolerability of sunitinib malate (Sutent) will be examined in previously untreated elderly patients (>70 years old) felt not to be candidates for standard cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Has measurable, metastatic NSCLC, other elderly NSCLC patients over 70 years of age who are not felt to be candidates for standard chemotherapy at the discretion of the treating physician may also be enrolled as long as they meet the criteria; these "special consideration" patients enrollment in the study must be approved by Dr. Reynolds or DR. Smith in Dr. Reynolds absence. Patients must have a nonsquamous histology to be eligible for this study.
* Has not received any prior chemotherapy for the current disease.
* Has an ECOG Performance status. Is 70 years of age or older.Has resolution of all acute toxic effects of radiotherapy or surgical procedures to NCI CTCAE.
* If fertile, patient (males only) has agreed to an acceptable method of birthcontrol to avoid pregnancy for the duration of the study and for a period of 2 months thereafter.
* Has signed the most recent Patient Informed Consent Form. Has signed a Pate int Authorization Form.

Exclusion Criteria:

* Has predominantly squamous NSCLC histology.
* Had prior treatment with study drugs or other drugs.
* Has a history of hypersensitivity to any component of the study drug. Has any evidence of an of antecedent hemoptysis, squamous histology, or ongoing anticoagulation or clotting diathesis.
* Pre-existing hemoptysis Grade 2, cavitating lesions or clear proximity or involvement of blood vessels.
* Has had major surgery or radiation therapy within 4 weeks of starting the study treatment.
* Has had NCI CTCAE (Version 3.0) Grade 3-4 hemorrhage within 4 weeks of starting the study treatment.
* Has a history of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan; however, treated, stable, and asymptomatic brain metastases are allowed.
* Has had any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism. Has ongoing cardiac dysrhythmias of NCI CTCAE (Version 3.0) Grade 2.
* Has prolonged QTc interval on baseline EKG. Has uncontrolled hypertension.
* Has pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Is receiving concurrent treatment on another clinical trial.
* Supportive care trials or non-treatment trials, (eg, QOL), are allowed.
* Is receiving concurrent immunotherapy, hormonal therapy, or radiation therapy.
* Is receiving concurrent investigational therapy or has received such therapy within the past 30 days.
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection.
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs.
* Is unable to comply with requirements of study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig H. Reynolds, MD, Principal Investigator — US Oncology Research, LLC; Ocala Oncology Center
Locations (13):
- United States (13):
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology - Arlington South, Arlington, Texas
  - Texas Oncology, P.A. - Bedford, Bedford, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 63
Completed | 29
Not Completed | 34
Not completed — Patient request | 11
Not completed — Hospitalized | 1
Not completed — Drug hold/delay more than 4 weeks | 1
Not completed — Adverse Event | 21

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 60
  Black | 1
  Hispanic | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Disease control rate = CR + PR + SD>=6-weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD) is defined as persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Every 6 weeks until progressive disease or death due to any cause, up to 36 month.
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 60
percentage of participants | 63.3 [49.9 to 75.4]

2. Secondary Outcome: Overall Response Rates (OR)
Description: Overall response rates = CR + PR. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 6 weeks until progressive disease or death due to any causes, up to 36 months.
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 60
percentage of participants | 6.7 [1.8 to 16.2]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from the date of registration to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at the date of last contact. Progressive disease (PD) is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: All patients were followed until progressive disease or death, up to 36 months.
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 63
months | 3.0 [0.1 to 25.1]

4. Secondary Outcome: 1-year Overall Survival (OS) Rate.
Description: OS is measured from the date of registration to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the date of last contact.
Time Frame: All patients were followed until death or up to 36 months.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants alive at 1yr
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 63
percentage of participants alive at 1yr | 26 [16 to 38]

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP is measured from the date of registration to the date of first documented disease progression or date of death due to progressive disease, whichever comes first. If a patient neither progresses nor dies due to progressive disease, this patient will be censored at the date of last contact. Progressive disease is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: All patients were followed until progressive disease or death, up to 36 months.
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 63
months | 4.5 [0.1 to 25.1]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 11/60
Other Adverse Events (participants affected / at risk) | 45/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=60)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ANEMIA HEMOLYTIC (NOS) (Blood and lymphatic system disorders) | 1 (1)
APPETITE DECREASED (Gastrointestinal disorders) | 2 (2)
BLEEDING GASTROINTESTINAL (Gastrointestinal disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (4)
DIVERTICULITIS (Infections and infestations) | 1 (1)
FATIGUE (General disorders) | 2 (2)
HEMORRHAGE (NOS) (Blood and lymphatic system disorders) | 1 (1)
JAUNDICE (Gastrointestinal disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1)
PAIN HEAD (General disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=60)
ANEMIA (Blood and lymphatic system disorders) | 5 (7)
ANOREXIA (Gastrointestinal disorders) | 13 (23)
CONSTIPATION (Gastrointestinal disorders) | 8 (11)
DEHYDRATION (Gastrointestinal disorders) | 4 (5)
DIARRHEA (Gastrointestinal disorders) | 18 (26)
DYSGUESIA (Gastrointestinal disorders) | 8 (8)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 (3)
FATIGUE (General disorders) | 26 (53)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 4 (4)
HEADACHE (General disorders) | 3 (3)
INFECTION FUNGAL (Infections and infestations) | 4 (5)
INSOMNIA (General disorders) | 3 (4)
MUCOSITIS (Infections and infestations) | 14 (20)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (5)
NAUSEA (Gastrointestinal disorders) | 14 (19)
NEUROPATHY (Nervous system disorders) | 4 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 9 (11)
PAIN MOUTH (Gastrointestinal disorders) | 3 (4)
PROTEINURIA (Renal and urinary disorders) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 (24)
VOMITING (Gastrointestinal disorders) | 8 (12)
WEAKNESS (General disorders) | 6 (7)
WEIGHT LOSS (General disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No